CLINICAL TRIAL: NCT00875628
Title: A Phase 1, Randomized, Double Blind (Sponsor-Open), Placebo Controlled, Dose Escalation, Multiple Dose Study To Investigate Safety, Tolerability, And Pharmacokinetics Of PF-00868554 In Japanese Healthy Adult Volunteers
Brief Title: A Study To Investigate Safety, Tolerability, And Pharmacokinetics Of PF-00868554 In Japanese Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A8121018
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Volunteers
Keywords: Japanese Healthy volunteers HCV pharmacokinetics PF-00868554 filibuvir
MeSH Terms: interventions — filibuvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Other): PF-00868554 100 mg or placebo
  Interventions: Drug: PF-00868554 or Placebo
- Cohort 2 (Other): PF-00868554 300 mg or placebo
  Interventions: Drug: PF-00868554 or Placebo
- Cohort 3 (Other): PF-00868554 600 mg or placebo
  Interventions: Drug: PF-00868554 or Placebo

INTERVENTIONS:
Drug: PF-00868554 or Placebo — Dosage Form: Oral solution Dosage: PF-00868554 100 mg or placebo under fasting conditions Frequency: BID (twice daily) Duration: 14 days
  Arms: Cohort 1
Drug: PF-00868554 or Placebo — Dosage Form: Oral solution Dosage: PF-00868554 300 mg or placebo under fasting conditions Frequency: BID (twice daily) Duration: 14 days
  Arms: Cohort 2
Drug: PF-00868554 or Placebo — Dosage Form: Tablet Dosage: PF-00868554 600 mg or placebo under fed conditions Frequency: BID (twice daily) Duration: 14 days
  Arms: Cohort 3

SUMMARY:
Investigation of safety, tolerability, and pharmacokinetics of PF-00868554 following multiple oral administrations of PF-00868554 in Japanese healthy adult volunteers.

DETAILED DESCRIPTION:
Study A8121018 was prematurely discontinued due to FDA instructions stating that Study A8121018 could not be performed under US IND 78,910, which was provided by the meeting on August 13, 2009. And then the termination was decided by Pfizer on September 8, 2009 prior to subject dosing with PF-00868554. There were no safety concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Japanese subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Male subjects with a history of subfertility/infertility and other conditions that in the opinion of the investigator may affect fertility.
* Exposure within the previous three months to a drug known to have a negative effect on skeletal muscle or reproductive organs.
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Plasma PF-00868554 concentrations | Day 1-Day 17
Urine PF-00868554 concentrations | Day 1 and Day 14
Adverse event monitoring and Physical examination | Day 0-Day 17
ECGs and vital signs (Blood pressure and Pulse rate) | Day 1-Day 17
Clinical safety laboratory tests | Day 0, Day 7, and Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121018&StudyName=A%20Study%20To%20Investigate%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20PF-00868554%20In%20Japanese%20Healthy%20Adult%20Volunteers